CLINICAL TRIAL: NCT00381836
Title: A Randomized, Multi-center Study to Assess the Effect of Darbepoetin Alfa (Aranesp®) for the Treatment of Anemia in Patients With Advanced Hormone Independent Prostate Cancer and Anaemia
Brief Title: Effect of Darbepoetin Alfa (Aranesp®) on Anemia in Patients With Advanced Hormone Independent Prostate Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Terminated by sponsor due to general risk that aranesp caused tumor progression
Sponsor: University of Aarhus (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2005-005658-37; LM: 2612-3148; Ethical: 20060074; Data Protection: 2005-41-6015
Record Dates: First submitted 2006-09-27; First posted 2006-09-28 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2008-02

CONDITIONS: Prostatic Neoplasms; Anemia
Keywords: Prostate Cancer; Anemia; Blood transfusion; Cancer; Critical illness; Drug efficacy; Drug safety; Drug tolerability; Erythropoietin; Fatigue; Hemoglobin; Human; Male; Multicenter study; Quality of life; Questionnaire; Randomized controlled trial; Recombinant erythropoietin
MeSH Terms: conditions — Prostatic Neoplasms; Anemia; Neoplasms; Critical Illness; Fatigue | interventions — Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Darbepoetin Alfa

SUMMARY:
The purpose of this study is to determine whether or not Aranesp® (Darbepoetin Alfa), administered every fourth week, is effective in the treatment of blood shortage (anemia) compared to standard care of treatment (blood transfusions) in patients with anemia due to hormone refractory prostate cancer.

DETAILED DESCRIPTION:
In the past, prostate cancer has been regarded a relatively benign disease, which elderly men were expected to die with rather than from, however, prostate cancer has become the second most common non-skin cancer in Danish men and the second most common cause of male cancer death. Two out of three patients with clinically significant prostate cancer die from and not with their cancer disease, and the misery of this population is evident. Regular treatments with opiates or equivalent drugs as well are required in nearly one third of the patients.

Patients with advanced hormone insensitive (refractory) prostate cancer have a median survival rate of about one year and during this time they often suffer from anemia due to reasons like blood loss, tumor infiltration of the bone marrow and even treatment with androgen deprivation. Compared to patients with other cancer types patients with prostate cancer have a significantly lower mean haemoglobin level. However, patients with hormone refractory prostate cancer have not previously been given much attention and the treatment of the frequent condition of chronic anemia in this group of patients seems casual. Therefore, Best Standard of Care (BSC) is defined as RBC transfusion if the hemoglobin is < 5,0 mmol/L (8,0 g/dl), and if there are signs or symptoms of anemia and supplemental iron if se-ferritin < 200 mcg/L.

Very little is known about erythropoietin treatment and quality of life in hormone refractory prostate cancer patients. A randomized Swedish study did investigate the influence of two different doses of epoetin beta on quality of life, hemoglobin level, need for red blood cell transfusion and safety, in the treatment of anemia in 180 patients suffering from advanced hormone-refractory prostate cancer. This study found the treatment to be safe and effective for the treatment in many of these patients. In many of these critically ill patients, the treatment improved quality of life and relieved fatigue symptoms.

Darbepoetin alpha (Aranesp®) is produced by gene-technology in Chinese Hamster Cells (CHO-K1). It has a biological effect and toxicity profile comparable to r-HuEPO; with the exception of a longer half-life which means that it can be administered less frequently without loosing clinical efficiency. Aranesp® has been well tolerated in studies conducted to this date. In this setting Aranesp® appears to be safe and well tolerated. Adverse events reported to date have generally been mild to moderate in severity and consistent with events and symptoms in cancer patients with chronic disease receiving chemotherapy (i.e. fatigue and gastrointestinal symptoms). Clinical studies have shown a higher frequency of thromboembolic reactions including deep vein thrombosis and pulmonary embolism in cancer patients receiving Aranesp therapy compared to patients receiving placebo. The clinical experience so far with Aranesp® has been published (15,16,17). Aranesp® is registered for clinical use in Europe and US.

Based on this the present study will evaluate the effect of Aranesp® on the haematopoietic response in patients with advanced hormone independent prostate cancer and anemia. Moreover, the effect of Aranesp® on quality of life, hemoglobin, necessity for RBC transfusion and hospital admissions, will be evaluated. The study will be performed as an open randomized trial. The use of r-HuEPO in cancer patients has been established and registered in other settings (as supportive treatment), and it has been shown that the preparation can be given without significant side effects. On the contrary, it is likely that patients may benefit from additional improvement in wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Male > 18 years
* Histologically proven prostate cell carcinoma
* Progression in PSA (10% elevation of nadir-value documented by two tests) at least 4 months after surgical orchiectomy or initiation of LHRH-agonist. Testosterone level must be below castration level
* All PSA values must be > 5 ng/ml
* Haemoglobin level below 11 g/dl (6.8 mmol/l)
* Haemoglobin level tested no later than 14 days prior to randomization
* A life expectancy of more than 3 months
* Participants must sign Informed consent according to local and national regulations and European Clinical Trial Directive

Exclusion Criteria:

* Known primary haematological disorder, which could cause anaemia
* Hypertension (diastolic blood pressure > 100 mmHg), refractory to treatment
* Symptomatic cardiovascular disease
* History of thromboembolic events during the last 12 months
* Concomitant Chemotherapy
* Active and severe liver disease
* Clinical significant inflammatory disease
* Concomitant or previous malignancies, which are likely to influence the treatment, evaluation and outcome of the current disease and therapy
* Concern of subject's compliance with the protocol procedures
* Previously included into the study
* Received erythropoietic therapy within 4 weeks before inclusion into the study
* Known positive antibody reaction to any erythropoietic agent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The haematopoietic response at week 4, 8, 12, 16 and 20

SECONDARY OUTCOMES:
Quality of Life (EQ-5D and QLQ-C30) at week 8 and 20
Number of blood transfusions at week 4, 8, 12, 16 and 20
Change in haemoglobin at week 4, 8, 12, 16 and 20
Number of days admitted to hospital during the 20 week study period

CONTACTS AND LOCATIONS:
Overall Officials: Michael Borre, MD, PhD, Principal Investigator — Department of Urology, Aarhus University Hospital
Locations (1):
- Department of Urology, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Background] Aus G, Hugosson J, Norlen L. Long-term survival and mortality in prostate cancer treated with noncurative intent. J Urol. 1995 Aug;154(2 Pt 1):460-5. doi: 10.1097/00005392-199508000-00033. PMID 7541864
- [Background] Potosky AL, Miller BA, Albertsen PC, Kramer BS. The role of increasing detection in the rising incidence of prostate cancer. JAMA. 1995 Feb 15;273(7):548-52. PMID 7530782
- [Background] Borre M, Nerstrom B, Overgaard J. The dilemma of prostate cancer--a growing human and economic burden irrespective of treatment strategies. Acta Oncol. 1997;36(7):681-7. doi: 10.3109/02841869709001337. PMID 9490083
- [Background] Brasso K, Friis S, Kjaer SK, Iversen P. [Prostatic cancer men under age 65. Occurrence and need for study]. Ugeskr Laeger. 1997 Apr 21;159(17):2543-5. Danish. PMID 9182383
- [Background] Borre M, Nerstrom B, Overgaard J. The natural history of prostate carcinoma based on a Danish population treated with no intent to cure. Cancer. 1997 Sep 1;80(5):917-28. PMID 9307192
- [Background] Aus G, Hugosson J, Norlen L. Need for hospital care and palliative treatment for prostate cancer treated with noncurative intent. J Urol. 1995 Aug;154(2 Pt 1):466-9. doi: 10.1097/00005392-199508000-00034. PMID 7541865
- [Background] Otnes B, Harvei S, Fossa SD. The burden of prostate cancer from diagnosis until death. Br J Urol. 1995 Nov;76(5):587-94. doi: 10.1111/j.1464-410x.1995.tb07783.x. PMID 8535677
- [Background] Carlsson P, Hjertberg H, Jonsson B, Varenhorst E. The cost of prostatic cancer in a defined population. Scand J Urol Nephrol. 1989;23(2):93-6. doi: 10.3109/00365598909180819. PMID 2787931
- [Background] Brasso K, Friis S, Juel K, Jorgensen T, Iversen P. The need for hospital care of patients with clinically localized prostate cancer managed by noncurative intent: a population based registry study. J Urol. 2000 Apr;163(4):1150-4. PMID 10737485
- [Background] Strum SB, McDermed JE, Scholz MC, Johnson H, Tisman G. Anaemia associated with androgen deprivation in patients with prostate cancer receiving combined hormone blockade. Br J Urol. 1997 Jun;79(6):933-41. doi: 10.1046/j.1464-410x.1997.00234.x. PMID 9202563
- [Background] Ornstein DK, Beiser JA, Andriole GL. Anaemia in men receiving combined finasteride and flutamide therapy for advanced prostate cancer. BJU Int. 1999 Jan;83(1):43-6. doi: 10.1046/j.1464-410x.1999.00844.x. PMID 10233450
- [Background] Johansson JE, Wersall P, Brandberg Y, Andersson SO, Nordstrom L; EPO-Study Group. Efficacy of epoetin beta on hemoglobin, quality of life, and transfusion needs in patients with anemia due to hormone-refractory prostate cancer--a randomized study. Scand J Urol Nephrol. 2001 Sep;35(4):288-94. doi: 10.1080/003655901750425864. PMID 11676354
- [Background] Dunn A, Carter J, Carter H. Anemia at the end of life: prevalence, significance, and causes in patients receiving palliative care. J Pain Symptom Manage. 2003 Dec;26(6):1132-9. doi: 10.1016/j.jpainsymman.2003.04.001. PMID 14654265
- [Background] Egrie JC, Browne JK. Development and characterization of novel erythropoiesis stimulating protein (NESP). Br J Cancer. 2001 Apr;84 Suppl 1(Suppl 1):3-10. doi: 10.1054/bjoc.2001.1746. PMID 11308268
- [Background] Heatherington AC, Schuller J, Mercer AJ. Pharmacokinetics of novel erythropoiesis stimulating protein (NESP) in cancer patients: preliminary report. Br J Cancer. 2001 Apr;84 Suppl 1(Suppl 1):11-6. doi: 10.1054/bjoc.2001.1747. PMID 11308269
- [Background] Glaspy J, Jadeja JS, Justice G, Kessler J, Richards D, Schwartzberg L, Rigas J, Kuter D, Harmon D, Prow D, Demetri G, Gordon D, Arseneau J, Saven A, Hynes H, Boccia R, O'Byrne J, Colowick AB. A dose-finding and safety study of novel erythropoiesis stimulating protein (NESP) for the treatment of anaemia in patients receiving multicycle chemotherapy. Br J Cancer. 2001 Apr;84 Suppl 1(Suppl 1):17-23. doi: 10.1054/bjoc.2001.1748. PMID 11308270
- [Background] Smith RE Jr, Tchekmedyian NS, Chan D, Meza LA, Northfelt DW, Patel R, Austin M, Colowick AB, Rossi G, Glaspy J. A dose- and schedule-finding study of darbepoetin alpha for the treatment of chronic anaemia of cancer. Br J Cancer. 2003 Jun 16;88(12):1851-8. doi: 10.1038/sj.bjc.6600994. PMID 12799626
- [Background] Bohlius J, Langensiepen S, Schwarzer G, Seidenfeld J, Piper M, Bennet C, Engert A. Erythropoietin for patients with malignant disease. Cochrane Database Syst Rev. 2004;(3):CD003407. doi: 10.1002/14651858.CD003407.pub2. PMID 15266483
- [Background] Bohlius J, Langensiepen S, Schwarzer G, Seidenfeld J, Piper M, Bennett C, Engert A. Recombinant human erythropoietin and overall survival in cancer patients: results of a comprehensive meta-analysis. J Natl Cancer Inst. 2005 Apr 6;97(7):489-98. doi: 10.1093/jnci/dji087. PMID 15812074
- [Background] Bohlius J, Wilson J, Seidenfeld J, Piper M, Schwarzer G, Sandercock J, Trelle S, Weingart O, Bayliss S, Djulbegovic B, Bennett CL, Langensiepen S, Hyde C, Engert A. Recombinant human erythropoietins and cancer patients: updated meta-analysis of 57 studies including 9353 patients. J Natl Cancer Inst. 2006 May 17;98(10):708-14. doi: 10.1093/jnci/djj189. PMID 16705125
- [Background] Williams KJ, Parker CA, Stratford IJ. Exogenous and endogenous markers of tumour oxygenation status: definitive markers of tumour hypoxia? Adv Exp Med Biol. 2005;566:285-94. doi: 10.1007/0-387-26206-7_38. PMID 16594164
- [Background] Varlotto J, Stevenson MA. Anemia, tumor hypoxemia, and the cancer patient. Int J Radiat Oncol Biol Phys. 2005 Sep 1;63(1):25-36. doi: 10.1016/j.ijrobp.2005.04.049. PMID 16111569